CLINICAL TRIAL: NCT01866904
Title: TIGRIS: Long-Term rIsk, Clinical manaGement and Healthcare Resource Utilization of Stable Coronary Artery dISease in Post Myocardial Infarction Patients
Brief Title: Long-Term rIsk, Clinical manaGement and Healthcare Resource Utilization of Stable CAD in Post MI Patients
Acronym: TIGRIS
Status: Terminated | Type: Observational
Why Stopped: Study was terminated in order to secure the data quality of the study in terms of follow-up rates and data completeness.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CMC-DUM-2013/1
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Stable Coronary Artery Disease (CAD), Myocardial Infarction
Keywords: Coronary artery disease, Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease, Autosomal Dominant, 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stable CAD patients aged 50 years or older: Stable CAD patients aged 50 years or older with documented history of presumed spontaneous MI with their most recent MI occurring 1 to 3 years prior to enrollment and have at least 1 additional risk factor

SUMMARY:
THis study is intended to provide contemporary data on the burden of disease in patients 1 to 3 years post-MI, including a description of patient characteristics, current treatment patterns, rate of major CV events, and healthcare resource utilization in a 'real world' patient population at high atherothrombotic risk.

DETAILED DESCRIPTION:
TIGRIS is a multinational, multi-centre, observational, prospective, longitudinal cohort study which will include stable CAD patients with history of MI 1-3 years ago and high risk of developing atherothrombotic events in a real world setting. The follow-up period is 3 years.

Patients will undergo clinical assessments and receive standard medical care as determined by the treating physician. Patients will not receive experimental intervention or experimental treatment as a consequence of their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

- Stable CAD patients aged 50 years or older with documented history of presumed spontaneous MI with their most recent MI occurring 1 to 3 years prior to enrollment and have at least 1 of the following risk factors: age ≥ 65 years; diabetes mellitus requiring medication; documented history of a second prior presumed spontaneous MI (>1 year ago); documented history of angiographic evidence of multivessel coronary artery disease; chronic renal dysfunction.

Exclusion Criteria:

* Presence of serious co-morbidities in the opinion of the investigator which may limit life expectancy (<1 year)
* Current participation in a blinded randomized clinical trial.
* Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient
* Patients receiving treatment of ticagrelor beyond 12 months, or off label use of ticagrelor.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable CAD patients aged 50 years or older with documented history of presumed spontaneous MI with their most recent MI occurring 1 to 3 years prior to enrollment and at least one additional risk factor for atherothrombotic events
Sampling Method: Probability Sample
Enrollment: 9284 (Actual)
Dates: Start 2013-06-19 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
MI, unstable angina with urgent revascularization, stroke, and death for any cause | in a 3-year follow-up period
  Event rates (time to first occurrence of any event from the composite of MI, unstable angina with urgent revascularization, stroke or death for any cause) in a three-year follow-up period.
Healthcare resource utilization | in a 3-year follow-up period
  Healthcare resource utilization associated with the events (MI, unstable angina with urgent revascularization, stroke or death for any cause) in a three-year follow-up period.

SECONDARY OUTCOMES:
Ischemic events (MI, unstable angina with urgent revascularization, ischemic stroke, CV death or death with unknown reason) | in a 3-year follow-up period
  To describe the rate of ischemic events (time to first occurrence of any event from the composite of MI, unstable angina with urgent revascularization, ischemic stroke, CV death or death with unknown reason) in a three-year follow-up period.
Bleeding events which require medical attention | in a 3 year follow-up period
  To describe the rate of bleeding events requiring medical attention.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zhang, M.D., PhD, Study Chair — AstraZeneca GMA; David Brieger, MBBS, PhD, Principal Investigator — Concord Repatriation General Hospital
Locations (309):
- United States (34):
  - Research Site, Huntsville, Alabama
  - Research Site, Los Angeles, California
  - Research Site, Santa Ana, California
  - Research Site, Torrance, California
  - Research Site, Ventura, California
  - Research Site, Clearwater, Florida
  - Research Site, Miami, Florida
  - Research Site, Tallahassee, Florida
  - Research Site, Tucker, Georgia
  - Research Site, Arlington Heights, Illinois
  - Research Site, Englewood, Illinois
  - Research Site, Lebanon, Indiana
  - Research Site, Auburn, Maine
  - Research Site, Bangor, Maine
  - Research Site, Columbia, Maryland
  - Research Site, Jackson, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Manhasset, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Sandusky, Ohio
  - Research Site, Abington, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Jackson, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Plano, Texas
  - Research Site, Burlington, Vermont
  - Research Site, Falls Church, Virginia
  - Research Site, Manassas, Virginia
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
- Argentina (6):
  - Research Site, Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Mendoza
  - Research Site, Salta
  - Research Site, Santa Fe
- Australia (16):
  - Research Site, Coffs Harbour, New South Wales
  - Research Site, Concord, New South Wales
  - Research Site, Kogarh, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, Newcastele, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Wollongong, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, Nambour, Queensland
  - Research Site, Southport, Queensland
  - Research Site, Woolloongabba, Queensland
  - Research Site, Epping, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Richmond, Victoria
  - Research Site, Fremantle, Western Australia
  - Research Site, Nedlands, Western Australia
- Belgium (10):
  - Research Site, Aalst
  - Research Site, Bonheiden
  - Research Site, Brasschaat
  - Research Site, Brussels
  - Research Site, Genk
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Ostend
  - Research Site, Overpelt
  - Research Site, Veurne
- Brazil (4):
  - Research Site, Campo Grande, Mato Grosso do Sul
  - Research Site, Blumenal, Santa Cantarina
  - Research Site, Marília, São Paulo
  - Research Site, São José do Rio Preto, São Paulo
- Canada (14):
  - Research Site, Saint John, New Brunswick
  - Research Site, Brampton, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Jérôme, Quebec
  - Research Site, Thetford-Mines, Quebec
  - Research Site, Québec
- China (15):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Lanzhou, Gansu
  - Research Site, Guangzhou, Guangdong
  - Research Site, Nanjing, Jiangsu
  - Research Site, Wuxi, Jiangsu
  - Research Site, Zhenjiang, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Jinzhou, Liaoning
  - Research Site, Jinan, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xian, Shanxi
  - Research Site, Taiyuan, Shanyuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Kunming, Yunnan
- Colombia (6):
  - Research Site, Medellín, Antioquia
  - Research Site, Barranquilla, Atlántico
  - Research Site, Cartagena, Caldas Department
  - Research Site, Manizales, Caldas Department
  - Research Site, Bucaramanga, Santander Dept
  - Research Site, Cali, Valle del Cauca Department
- Denmark (8):
  - Research Site, Aalborg
  - Research Site, Arhus N
  - Research Site, Copenhagen
  - Research Site, Haderslev
  - Research Site, Hellerup
  - Research Site, København NV
  - Research Site, København S
  - Research Site, Randers
- Finland (4):
  - Research Site, Jyväskylä
  - Research Site, Rovaniemi
  - Research Site, Tampere
  - Research Site, Turku
- France (16):
  - Research Site, Abbeville
  - Research Site, Arras
  - Research Site, Boulogne-Billancourt
  - Research Site, Briis Sous Forge
  - Research Site, Corbeille Essone
  - Research Site, Dijon
  - Research Site, La Rochelle
  - Research Site, Langres
  - Research Site, Le Chesnay
  - Research Site, Le Coudray
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Nice
  - Research Site, Roubaix
  - Research Site, Salouël
  - Research Site, Toulouse
- Germany (28):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Chemnitz
  - Research Site, Cloppenburg
  - Research Site, Coburg
  - Research Site, Cologne
  - Research Site, Dresden
  - Research Site, Erfurt
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Frankfurt M
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Koblenz
  - Research Site, Leipzig
  - Research Site, Leverkusen
  - Research Site, Ludwigshafen
  - Research Site, Lübeck
  - Research Site, Mainz
  - Research Site, Merseburg
  - Research Site, Mönchengladbach
  - Research Site, München
  - Research Site, Potsdam
  - Research Site, Soltau
  - Research Site, Stuttgart
  - Research Site, Ulm
- India (15):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Surat, Gujarat
  - Research Site, Bangalore, Karnataka
  - Research Site, Thrisur, Kerala
  - Research Site, Trivandrum, Kerala
  - Research Site, Indore, Madhya Pradesh
  - Research Site, Mumbai, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Mohali, Punjab
  - Research Site, Jaipur, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Noida, Uttar Pradesh
  - Research Site, Kolkata, West Bengal
- Italy (14):
  - Research Site, Ancona
  - Research Site, Bologna
  - Research Site, Catania
  - Research Site, Lagosanto FE
  - Research Site, Lido di Camaiore
  - Research Site, Massa Carrara
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Nuoro
  - Research Site, Palermo
  - Research Site, Perugia
  - Research Site, Prato
  - Research Site, Sassari
  - Research Site, Treviso
- Japan (31):
  - Research Site, Toyoake-shi, Aichi-ken
  - Research Site, Chiba, Chiba
  - Research Site, Kisarazu-shi, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukui-shi, Fukui
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Kurume-shi, Fukuoka
  - Research Site, Maebashi, Gunma
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tomakomai-shi, Hokkaido
  - Research Site, Amagasaki-shi, Hyōgo
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Morioka, Iwate
  - Research Site, Isehara-shi, Kanagawa
  - Research Site, Sagamihara-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kochi, Kochi
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Sendai, Miyagi
  - Research Site, Tenri-shi, Nara
  - Research Site, Hirakata-shi, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Suita-shi, Osaka
  - Research Site, Kusatsu-shi, Shiga
  - Research Site, Izunokuni-shi, Shizuoka
  - Research Site, Shizuoka, Shizuoka
  - Research Site, Komatsujima-shi, Tokushima
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Chuo-Ku, Tokyo
  - Research Site, Wakayama, Wakayama
- Mexico (10):
  - Research Site, Torreón, Coahuila
  - Research Site, Tijuana, Estado de Baja California
  - Research Site, Guadalajara, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Querétaro City, Querétaro
  - Research Site, Toluca, State of Mexico
  - Research Site, Chihuahua City
  - Research Site, Oaxaca City
  - Research Site, Puebla City
  - Research Site, San Luis Potosí City
- Netherlands (17):
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Blaricum
  - Research Site, Delft
  - Research Site, Doetinchem
  - Research Site, Ede
  - Research Site, Groningen
  - Research Site, Haarlem
  - Research Site, Hardenberg
  - Research Site, Heerlen
  - Research Site, Hoofddorp
  - Research Site, Hoogeveen
  - Research Site, IJssel
  - Research Site, Meppel
  - Research Site, Sittard-Geleen
  - Research Site, The Hague
  - Research Site, Zutphen
- Norway (3):
  - Research Site, Fredrikstad
  - Research Site, Oslo
  - Research Site, Stavanger
- Portugal (8):
  - Research Site, Braga
  - Research Site, Canelas
  - Research Site, Faro
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Senhora da Hora
  - Research Site, Setúbal
  - Research Site, Viana do Castelo
- Romania (11):
  - Research Site, Arad
  - Research Site, Brăila
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Drobeta-Turnu Severin
  - Research Site, Focşani
  - Research Site, Piteşti
  - Research Site, Sibiu
  - Research Site, Slatina
  - Research Site, Timișoara
- South Korea (9):
  - Research Site, Chungcheongbuk-do, Cheongju-si
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Jinju, Gyeongsangnam-do
  - Research Site, Jeonju, Jeollabuk-do
  - Research Site, Gwangju, Jeollanam-do
  - Research Site, Daejeon, Jung-gu
  - Research Site, Daegu, Nam-gu
  - Research Site, Busan, Seo-gu
  - Research Site, Seoul, Sudogwon
- Spain (14):
  - Research Site, Seville, Andalusia
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Toledo, Castille-La Mancha
  - Research Site, Barcelona, Catalonia
  - Research Site, Vic, Catalonia
  - Research Site, Cáceres, Extremadura
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Baza, Granada
  - Research Site, Alicante
  - Research Site, Almería
  - Research Site, Granada
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Murcia
- Turkey (Türkiye) (6):
  - Research Site, Ankara
  - Research Site, Aydin
  - Research Site, Diyarbak?r
  - Research Site, Istanbul
  - Research Site, Merkez
  - Research Site, Mersin
- United Kingdom (8):
  - Research Site, Airdrie
  - Research Site, Cambridge
  - Research Site, East Kilbride
  - Research Site, London
  - Research Site, Portadown
  - Research Site, Sheffield
  - Research Site, Taunton
  - Research Site, Wolverhampton
- Venezuela (2):
  - Research Site, Valencia, Carabobo
  - Research Site, Caracas, Miranda

REFERENCES:
- [Derived] Krishnamurthy SN, Pocock S, Kaul P, Owen R, Goodman SG, Granger CB, Nicolau JC, Simon T, Westermann D, Yasuda S, Andersson K, Brandrup-Wognsen G, Hunt PR, Brieger DB, Cohen MG. Comparing the long-term outcomes in chronic coronary syndrome patients with prior ST-segment and non-ST-segment elevation myocardial infarction: findings from the TIGRIS registry. BMJ Open. 2023 Dec 18;13(12):e070237. doi: 10.1136/bmjopen-2022-070237. PMID 38110389
- [Derived] Nicolau JC, Owen R, Furtado RHM, Goodman SG, Granger CB, Cohen MG, Westermann D, Yasuda S, Simon T, Hedman K, Hunt PR, Brieger DB, Pocock SJ. Long-term outcomes among stable post-acute myocardial infarction patients living in rural versus urban areas: insights from the prospective, observational TIGRIS registry. Open Heart. 2023 Aug;10(2):e002326. doi: 10.1136/openhrt-2023-002326. PMID 37604649
- [Derived] Bagai A, Ali FM, Gregson J, Alexander KP, Cohen MG, Sundell KA, Simon T, Westermann D, Yasuda S, Brieger D, Goodman SG, Nicolau JC, Granger CB, Pocock S. Multimorbidity, functional impairment, and mortality in older patients stable after prior acute myocardial infarction: Insights from the TIGRIS registry. Clin Cardiol. 2022 Dec;45(12):1277-1286. doi: 10.1002/clc.23915. Epub 2022 Nov 1. PMID 36317424
- [Derived] Carnicelli AP, Owen R, Pocock SJ, Brieger DB, Yasuda S, Nicolau JC, Goodman SG, Cohen MG, Simon T, Westermann D, Hedman K, Andersson Sundell K, Granger CB. Atrial fibrillation and clinical outcomes 1 to 3 years after myocardial infarction. Open Heart. 2021 Dec;8(2):e001726. doi: 10.1136/openhrt-2021-001726. PMID 34911791
- [Derived] Russo JJ, Yan AT, Pocock SJ, Brieger D, Owen R, Sundell KA, Bagai A, Granger CB, Cohen MG, Yasuda S, Nicolau JC, Brandrup-Wognsen G, Westermann D, Simon T, Goodman SG. Determinants of long-term dual antiplatelet therapy use in post myocardial infarction patients: Insights from the TIGRIS registry. J Cardiol. 2022 Apr;79(4):522-529. doi: 10.1016/j.jjcc.2021.10.024. Epub 2021 Nov 29. PMID 34857432
- [Derived] Pocock S, Brieger DB, Owen R, Chen J, Cohen MG, Goodman S, Granger CB, Nicolau JC, Simon T, Westermann D, Yasuda S, Hedman K, Mellstrom C, Andersson Sundell K, Grieve R. Health-related quality of life 1-3 years post-myocardial infarction: its impact on prognosis. Open Heart. 2021 Feb;8(1):e001499. doi: 10.1136/openhrt-2020-001499. PMID 33563776
- [Derived] Nicolau JC, Brieger D, Owen R, Furtado RHM, Goodman SG, Cohen MG, Simon T, Westermann D, Granger CB, Grieve R, Yasuda S, Chen J, Hedman K, Mellstrom C, Brandrup-Wognsen G, Pocock SJ. Diabetes association with self-reported health, resource utilization, and prognosis post-myocardial infarction. Clin Cardiol. 2020 Dec;43(12):1352-1361. doi: 10.1002/clc.23476. Epub 2020 Nov 4. PMID 33146924
- [Derived] Westermann D, Goodman SG, Nicolau JC, Requena G, Maguire A, Chen JY, Granger CB, Grieve R, Pocock SJ, Blankenberg S, Vega AM, Yasuda S, Simon T, Brieger D; TIGRIS Study Investigators. Rationale and design of the long-Term rIsk, clinical manaGement, and healthcare Resource utilization of stable coronary artery dISease in post-myocardial infarction patients (TIGRIS) study. Clin Cardiol. 2017 Dec;40(12):1197-1204. doi: 10.1002/clc.22837. Epub 2017 Dec 16. PMID 29247524
- [Derived] Goodman SG, Nicolau JC, Requena G, Maguire A, Blankenberg S, Chen JY, Granger CB, Grieve R, Pocock SJ, Simon T, Yasuda S, Vega AM, Brieger D; TIGRIS Study Investigators. Longer-term oral antiplatelet use in stable post-myocardial infarction patients: Insights from the long Term rIsk, clinical manaGement and healthcare Resource utilization of stable coronary artery dISease (TIGRIS) observational study. Int J Cardiol. 2017 Jun 1;236:54-60. doi: 10.1016/j.ijcard.2017.02.062. Epub 2017 Feb 21. PMID 28268087
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1822&filename=TIGRIS_CSR_%20synopsis_final_Redacted.pdf